CLINICAL TRIAL: NCT00645931
Title: Proposal for a Bone Marrow Transplant Pre, Post, and Long Term Psychological Evaluation Study.
Brief Title: Psychological Effects of Bone Marrow Transplants in Children
Status: Completed | Type: Observational
Sponsor: Corewell Health West (Other)
Collaborators: Helen DeVos Children's Hospital (Other)
Responsible Party: Heather L Hammerstrom, Spectrum Health
Other Study IDs: 2004-105; 2004-105
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Psychological
Keywords: Bone Marrow; Bone Marrow Transplant; Pediatric; Psychological Impact; Psychology
MeSH Terms: interventions — Proteins; Caloric Restriction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: protein and calorie controlled diet and self-hypnotic relaxation — daily

SUMMARY:
This study is designed to examine the psychological effects of bone marrow transplants on children and their families. The investigators hypothesis is that families who show signs of psychological distress before transplant will continue those signs post transplant. The investigators are examining cognitive placement, emotional placement and other psychological factors in both the child undergoing transplant and his or her parent.

DETAILED DESCRIPTION:
Previous research on bone marrow transplants has conflicting results concerning the effects of maladjustment. The current research is conducted in consortium with DeVos Children's Hospital. Children receiving bone marrow transplants are assessed using the Child Behavior Check List (CBCL) and Cognitive based testing. Parents are assessed using the Parenting Stress Index (PSI). Children and parents are evaluated prior to transplant and then 50 days, 6 months, and one year post transplant. Descriptive statistics are currently being used to determine results.

ELIGIBILITY:
Inclusion Criteria:

* bone marrow transplant eligible patients
* 18 years and under
* male and female

Exclusion Criteria:

* over the age of 18

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients under the age of 18
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2004-06; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The specific measure that will be used to determine the effect of the intervention(s). The description should included the time at which the measure will be taken. Examples: all cause mortality at one year; score on a depression rating scale at 6 weeks | 1 year post transplant

SECONDARY OUTCOMES:
Other measures that will be used to evaluate the intervention(s), and that are specified in the protocol. The description should include the time at which the measures will be taken. Ex. cardiovascular mortality at 6 mos.; functional status at 4 wks | 1 year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hammerstrom, BA, Principal Investigator — Helen DeVos Children's Hospital
Locations (1):
- Helen DeVos Children's Hospital, Grand Rapids, Michigan, United States